CLINICAL TRIAL: NCT04307511
Title: A Randomized Controlled sTudy of Low Dose vs Standard Dose of tIcaGrelor on Platelet Function After intErvention for Acute Coronary syndRome in Diabetes Mellitus Patients
Brief Title: A sTudy of Low Dose vs Standard Dose of tIcaGrelor on Platelet Function After intErvention for Acute Coronary syndRome in Diabetes Mellitus Patients
Acronym: TIGER-diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Principal Investigator, Hou Lei, Clinical Professor, Shanghai Tong Ren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020PYN
Record Dates: First submitted 2020-03-08; First posted 2020-03-13 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Acute Coronary Syndrome Patients With Diabetes After PCI
MeSH Terms: interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose DAPT therapy (Experimental): treated with ticagrelor 60mg plus aspirin 100 mg for 11 months after one month standard DAPT(ticagrelor 90mg plus aspirin 100 mg )treatment
  Interventions: Drug: Ticagrelor; Drug: Aspirin
- standard dose DAPT therapy (Active Comparator): treated with ticagrelor 90mg and aspirin 100mg after PCI for 12 months as the standard group
  Interventions: Drug: Ticagrelor; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor — 60mg ticagrelor based DAPT vs 90mg ticagrelor based DAPT vs 90mg ticagrelor monotherapy
Drug: Aspirin — Aspirin

SUMMARY:
In this study, the investigates try to confirm the hypothesis that low dose ticagrelor(60mg) had similar anti-platelets function compared with the standard dose ticagrelor in acute coronary syndrome patients with diabetes. Totally 40 ACS patients with diabetes will be divided into 2 groups randomly after PCI for one month. Group 1 will be treated with ticagrelor 90mg and aspirin 100mg after PCI for 12 months as the standard group; Group2 will be treated with ticagrelor 60mg plus aspirin 100 mg for 11 months after one month standard DAPT treatment. The platelets function will be tested in VASP and TEG methods at 1 and 2 months after PCI as the primary endpoints.The clinical events will be observed 12 months after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age and less than 90 years old
2. Patients should have undergone successful percutaneous coronary intervention with drug-eluting stent for acute coronary syndrome with diabetes mellitus.
3. Subject understand the study requirements and the treatment procedures and
4. provided informed consent before the procedure

Exclusion Criteria:

1. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
2. Active bleeding
3. Known hypersensitivity or contraindication to study medications
4. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
5. Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment).
6. Subjects with Cerebral hemorrhage history
7. Subjects with stroke history in half a year
8. subjects with active malignant tumor
9. subjects with whom oral anticoagulants are needed
10. Other conditions which the investigators think not applicable to the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
changes of PRI detected by VASP | changes of PRI from baseline (1 months after index PCI) to 2 months after index PCI
  platelet reactivity index (PRI) detected by VASP (Vasodilator Stimulated Phosphoprotein) Phosphoprotein)
changes of Maximum Amplitude (MA) detected by TEG | changes of MA from baseline (1 months after index PCI) to 2 months after index PCI
  Maximum Amplitude (MA) detected by TEG(Thromboelastography)

CONTACTS AND LOCATIONS:
Locations (1):
- shanghai Tongren hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No